CLINICAL TRIAL: NCT03025295
Title: The Effect of Orexin on Delayed Emergence of General Anesthesia in Dexmedetomidine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: XZ2015020
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Anesthesia
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Induction dose of dexmedetomidine is 1ug/kg with 10min, maintain dose is 0.4ug/kg/h until 30 min before surgery completion.
  Interventions: Drug: Dexmedetomidine
- Saline group (Placebo Comparator): Control group given equal volume of saline with the dexmedetomidine group.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine is common used to improve the prognosis and life quality of patients.
  Other Names: Dexmedetomidine is a highly selective α2-adrenoceptor agonist.
  Arms: Dexmedetomidine group
Drug: Saline — It is safe Placebo.
  Other Names: It is safe Placebo.
  Arms: Saline group

SUMMARY:
The current study is designed to investigate the difference of plasma orexin A levels between Dexmedetomidine group and controlled group at emergence time from total intravenous anesthesia who will undergo elective lumbar surgery.

DETAILED DESCRIPTION:
DESIGNING: Fifty-one patients with ASA physical status I or II scheduled for elective surgery under general anesthesia (lasting for 2h to 4h) were enrolled. Anesthesia was induced with propofol 1-2mg/kg and sufentanyl 0.2-0.3μg/kg. Following muscle relaxation with iv cisatracurium besylate 0.2mg/kg endotracheal intubation was performed. Anesthesia was maintained with target controlled infusion propofol (targeted concentration:2-5ug/ml ) and remifentanil (targeted concentration: 2-6ng/ml ). Muscle relaxation was maintained with intermittent, but it do not injected in 1h before surgery completion. Propofol and remifentanil were titrated to maintain the bispectral index (BIS) between 40 and 60 during anesthesia. The end-tidal carbon dioxide level was maintained between 30 and 40 mmHg by controlled mechanical ventilation. When the surgery was completed the investigators adjust the targeted concentration of propofol 2ug/ml and targeted concentration of remifentanil to 2ng/ml then stop all anesthetics. Dexmedetomidine group target controlled infusion dexmedetomidine (induction dose 1ug/kg with 10min, maintain dose 0.4ug/kg/h until 30min before surgery completion). Control group infusion same saline. Record time from stopping anesthetics to emergence and total doses of anesthetics. Arterial blood (2.5ml) was collected at the following time, such as before and 1h after induction of anesthesia, at emergence (1 min after tracheal extubation) and half an hour after tracheal extubation. 2.0ml Arterial blood was centrifuged at 3000 rpm for 15min at -4 ◦C in order to separate plasma then stored at -80 ◦C until assay for orexin A concentrations. 0.5ml Arterial blood was measured blood glucose.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is Adult (≥18 years old and ≤60 years old)
2. Participants with a Body Mass Index (BMI) 20-25 kg/m2
3. Participants with ASA physical status Ⅰor Ⅱ
4. Participants with Heart function rating Ⅰor Ⅱ
5. Patients will undergo elective surgery and general anesthesia
6. The operation time is 2h to 4h.

Exclusion Criteria:

1. Participant is a pregnant woman or a nursing mother.
2. Participants have a history of narcotics allergic reactions.
3. Indices of liver or kidney function is twice higher than normal.
4. Participants have a history or diagnosis of depression.
5. Participants have a history of Brain Trauma.
6. Participants have a history of narcotics addiction or drug addiction.
7. Participants or his family have an International Classification of Sleep
8. Disorders diagnosis of obstructive sleep apnea syndrome.
9. Patients are refuse this trail or are not able to sign informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
orexin A concentrations | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Zhihua Wang, M.D., Study Chair — General Hospital of Ningxia Medical University
Locations (1):
- Anesthesiology department of General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: Undecided